CLINICAL TRIAL: NCT05954598
Title: Effect of Probiotic vs Placebo on Cognition Outcomes in Patients With Bipolar Disorder: A Randomized Clinical Trial
Brief Title: Effect of Probiotic vs Placebo on Cognition Outcomes in Patients With Bipolar Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Hu ShaoHua, Professor, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIT20220105C-R1
Record Dates: First submitted 2023-07-04; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic (Experimental): The intervention group received 12 weeks of probiotic intervention from the beginning of the study,and at the start of the study at week 13, both groups received 12 consecutive weeks of probiotic intervention
  Interventions: Dietary Supplement: probiotic
- placebo (Placebo Comparator): The waiting group received 12 consecutive weeks of placebo intervention from the start of the study, and at the start of the study at week 13, both groups received 12 consecutive weeks of probiotic intervention
  Interventions: Dietary Supplement: probiotic

INTERVENTIONS:
Dietary Supplement: probiotic — This study was designed as a randomized double-blind controlled study. The enrolled subjects were randomized into two groups: intervention group and waiting intervention group. The intervention group received 12 weeks of probiotic intervention from the start of the study, and the waiting group received 12 weeks of placebo intervention from the start of the study. At the start of the study, both groups received 12 weeks of probiotic intervention.

SUMMARY:
Bipolar disorder has a high hospitalization rate, suicide rate and disability rate, and cognitive dysfunction is one of the core clinical symptoms of bipolar disorder. Cognitive recovery has become a new target and a new target for clinical treatment. In recent years, gut microbiome has been recognized as one of the neuropathological mechanisms of bipolar disorder. This study aims to study the effect of probiotics on cognitive function in stable bipolar disorder patients and the possible mechanism of action. A total of 100 patients with stable bipolar disorder were enrolled into the control group and the experimental group in a random double-blind way to evaluate the intestinal microecology, clinical symptom improvement, cognitive function and side effects before and after treatment between the two groups, and further explore the possible mechanism of action of the experimental drug.

DETAILED DESCRIPTION:
Bipolar disorder has a high hospitalization rate, suicide rate and disability rate, and cognitive dysfunction is one of the core clinical symptoms of bipolar disorder. Cognitive recovery has become a new target and a new target for clinical treatment. In recent years, gut microbiome has been recognized as one of the neuropathological mechanisms of bipolar disorder. This study aims to study the effect of probiotics on cognitive function in stable bipolar disorder patients and the possible mechanism of action. A total of 100 patients with stable bipolar disorder were enrolled into the control group and the experimental group in a random double-blind way. This study was designed as a randomized double-blind controlled study. The enrolled subjects were randomized into two groups: intervention group and waiting intervention group. The intervention group received 12 weeks of probiotic intervention from the start of the study, and the waiting group received 12 weeks of placebo intervention from the start of the study. At the start of the study, both groups received 12 weeks of probiotic intervention. This study to compare the dynamic changes of cognitive function and resting brain network in stable bipolar disorder patients before and after using probiotics, and to compare the changes of physical symptoms, sleep and serum cortisol levels in stable bipolar disorder patients before and after the use of probiotics between the two groups, and further explore the possible mechanism of action of the experimental drug.

ELIGIBILITY:
Inclusion Criteria：

1）Both biological parents were Han. 2) Age 16-65 years old, male or female; 3) The subjects met the DSM-5 clinical diagnostic criteria for bipolar disorder, and the 17-item Hamilton Depression Scale score (HAMD-17) ≤16 points, Hamilton Anxiety Scale score ≤7 points, and Young Mania Scale score ≤5 points were maintained for more than 2 months. All enrolled patients were evaluated by a professional and systematically trained psychiatrist.

4) No probiotic preparations such as yogurt were taken within 1 month before enrollment; 5) No clear history of respiratory tract, urinary system, digestive system infection or antibiotic use within 1 month before enrollment; 6) The drug regimen remained stable within 1 month before enrollment; 7) Perceived Deficits Questionnaire (PDQ) score ≥17 points; 8) Right-handed; 9) Primary school education or above; 10) Informed consent of patients and their families to this study. Exclusion Criteria：

1. Those who meet the DSM-5 diagnostic criteria for schizophrenia, depression, neurodevelopmental disorders, dementia, memory impairment, or other cognitive disabilities;
2. Those who had used ECT before enrollment;
3. Those who currently have serious suicidal thoughts or behaviors, or who are severely agitated;
4. Those who cannot follow the doctor's advice or have no guardian;
5. Pregnant or lactating women, or those planning pregnancy.
6. Patients with abnormal brain structure or any MRI contraindications found by magnetic resonance examination.
7. Mental disorders caused by substance abuse (alcohol, drugs, etc.), people with serious physical diseases, such as thyroid disease, heart disease, abnormal liver and kidney function, etc.; 8）Can not tolerate any probiotic preparations or have a history of allergy.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Scores change from Baseline the number symbol test at 24 weeks | week0，week8，week12，week24

SECONDARY OUTCOMES:
Visuospatial function | week0，week8，week12，week24
  Scores change from Baseline the short visuospatial memory test at 24 weeks
Working memory | week0，week8，week12，week24
  Scores change from Baseline the Spatial span test at 24 weeks
MRI (Functional connectivity, network features) | week0，week12，
  change from Baseline the Functional connectivity and network features at 12 weeks
Somatic symptoms | week0，week8，week12，week24
  change from Baseline the Somatic symptoms self-rating scale at 24 weeks，the minimum and maximum values：0-80， higher scores mean a worse outcome
Sleep | week0，week8，week12，week24
  change from Baseline the Sleep Quality Questionnaire (PSQI) at 24 weeks
Changes in serum cortisol levels | week0，week8，week12
  Changes from Baseline serum cortisol levels at 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine (FAHZU), Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No